CLINICAL TRIAL: NCT06515730
Title: RandomizEd compariSOn of Apixaban Versus Warfarin in Patients With Left VEntricular Thrombus After Acute Myocardial Infarction (RESOLVE-AMI)
Brief Title: Treatment With Apixaban Versus Warfarin in Patients With Left Ventricular Thrombus After Acute Myocardial Infarction
Acronym: RESOLVE-AMI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska Trial Alliance (Industry); Swedish Heart Lung Foundation (Other); The Swedish Research Council (Other Government); Stockholm County Council ALF/PPG (Unknown)
Responsible Party: Principal Investigator, Moa Simonsson, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RESOLVE-AMI
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-07

CONDITIONS: Left Ventricular Thrombus; Acute Myocardial Infarction
Keywords: Apixaban; warfarin
MeSH Terms: interventions — apixaban; Warfarin; Vitamin B 6

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, multicenter, open-label, blinded outcome assessment, parallel arm, active comparator, randomized study
Who Masked: Outcomes Assessor
Masking Description: Assessment of the primary outcome of thrombus resolution will be performed through review of images by researchers who are blinded to the treatment assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apixaban (Experimental): Apixaban 5 mg twice a day, reduced to 2.5 mg twice a day for participants with any 2 of following criteria: age > 80 years, serum creatinine > 133 μmol/L or body weight <60 kg. Participants with severe renal failure defined as creatinine clearance 15-29 ml/min/1.73 m2, should also receive the reduced dose of 2.5 mg twice a day.
  Interventions: Drug: Apixaban
- Warfarin (Active Comparator): Warfarin 2,5 mg once daily with individual dosing according to coagulation assays with an international normalized ratio (INR) goal of 2.0-3.0. Bridging with low-molecular-weight-heparin with a dose of dalteparin 200 units/kg but maximum 18 000 units or enoxaparin 150 units/kg, until therapeutic INR is recommended.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Apixaban — 5 mg tablet twice a daily with dose reduction according to label
  Other Names: Eliquis
  Arms: Apixaban
Drug: Warfarin — 2.5 mg tablet once daily, with individual dosing according to coagulation tests
  Other Names: Waran
  Arms: Warfarin

SUMMARY:
The optimal anticoagulant for the treatment of left ventricular (LV) thrombus following acute myocardial infarction (AMI) is unclear. The aim of this multicenter randomized study is to evaluate the efficacy of apixaban versus warfarin with respect to thrombus resolution in patients with LV thrombus after AMI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of signing the informed consent
* LV thrombus confirmed on TTE* day 1-28 after the AMI
* Signed informed consent
* Criteria applicable only for female subjects: Women of childbearing potential must provide a negative pregnancy test not be breastfeeding and be willing and able to use highly effective contraception. Women of non-childbearing potential must be 1 year post-menopausal.

Exclusion Criteria:

* Ongoing* treatment with anticoagulant therapy due to Mechanical heart valve prosthesis Atrial fibrillation with or without significant mitral valve stenosis Venous thromboembolism requiring anticoagulant therapy Thrombophilia requiring anticoagulant therapy Preexisting LV thrombus already treated with anticoagulant therapy Other reasons for anticoagulant therapy
* High bleeding risk Active non-trivial bleeding Known chronic bleeding disorder Severe anemia defined as hemoglobin < 80g/L Thrombocytopenia defined as platelet count < 80 x 10^9
* Known significant liver disease (e.g. acute hepatitis, chronic active hepatitis, cirrhosis) or known hepatic insufficiency classified as Child-Pugh C or D at randomization
* Known allergy, intolerance or hypersensitivity to either of the study interventions
* Any contraindication for the use of an anticoagulant or listed in the local labelling for apixaban or warfarin.
* Participation in other study investigating effects and safety of anticoagulant treatment.
* Known current alcohol or drug abuse
* Any other condition, as judged by the investigator, that would make the participant unsafe or unsuitable for the study or life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2028-04-08 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of participants with thrombus resolution at 3 months | 3 months
  Thrombus resolution will be evaluated on transthoracic echocardiogram (TTE*) at 3 months

SECONDARY OUTCOMES:
Clinically relevant bleeding at 3 and 12 months | 3 and 12 months
  Clinical relevant bleeding defined as Bleeding Academy Research Consortium (BARC) 2, 3 or 5 bleeding.
  The BARC bleeding scale ranges from 0 to 5, where 0 is equal to no bleeding, with increasing severity from 1 through 5, where 5 represents fatal bleeding. Major bleeding is most often defined as BARC 3 and 5. BARC 4 bleeding is coronary artery bypass grafting (CABG) related bleeding.
Severe bleeding at 3 and 12 months | 3 and 12 months
  Severe bleeding defined as BARC 3 or 5. For definition of the BARC bleeding scale please see Outcome 2 above.
Separate bleeding outcomes at 3 and 12 months | 3 and 12 months
  Separate bleeding outcomes defined as fatal, intracranial, gastro-intestinal uro-genital or other bleeding
Major adverse cardiovascular outcomes (MACE) at 3 and 12 months | 3 and 12 months
  MACE is defined as a composite of non-fatal myocardial infarction, non-fatal stroke or cardiovascular death
Stroke or systemic embolism at 3 and 12 months | 3 and 12 months
  Composite of ischemic stroke or systemic embolism
LV thrombus status at 12 months | 12 months
  Recurrence (or in absence of resolution of LV thrombus at 3 months, persistence) of LV thrombus on TTE at 12 months
Net adverse clinical outcomes | 3 and 12 months
  Composite of MACE and. BARC 2, 3 or 5 bleeding. For definition of MACE and BARC bleeding scale please see Outcome 2 and 5 above.

CONTACTS AND LOCATIONS:
Overall Officials: Moa Simonsson, MD, PhD, Principal Investigator — Department of Medicine Solna, Karolinska Institutet
Locations (16):
- Sweden (16):
  - Falu lasarett, Falun
  - Sahlgrenska University hospital, Mölndal, Gothenburg
  - Sahlgrenska University hospital, Östra, Gothenburg
  - Sahlgrenska University hospital, Gothenburg
  - Linköping University hospital, Linköping
  - Skånes Universitetssjukhus Lund, Lund
  - Skånes University hospital, Malmö, Malmo
  - Vrinnevi hospital, Nörrköping
  - Örebro University hospital, Örebro
  - Karolinska Insitutet, Stockholm
  - Danderyds hospital, Stockholm
  - Karolinska Univerity Hospital, Stockholm
  - Sankt Görans Hospital, Stockholm
  - Södersjukhuset, Stockholm
  - Uppsala Akademiska hospital, Uppsala
  - Västmanlands hospital, Västerås, Västerås

IPD SHARING:
Plan to Share IPD: No